CLINICAL TRIAL: NCT00302510
Title: Therapeutic Effect of Immunoadsorption for Patients With Lipoprotein
Brief Title: Therapeutic Effect of Immunoadsorption for Patients With Lipoprotein Glomerulopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0608
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2008-07

CONDITIONS: Treatment
Keywords: lipoprotein glomerulopathy; treatment; immunoadsorption; apolipoprotein E
MeSH Terms: conditions — Lipoprotein Glomerulopathy | interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immunoadsorption (Placebo Comparator)
  Interventions: Procedure: immunoadsorption

INTERVENTIONS:
Procedure: immunoadsorption — immunoadsorption

SUMMARY:
The purpose of this study is to assess the efficacy and safety of immunoadsorption in the treatment of lipoprotein glomerulopathy.

DETAILED DESCRIPTION:
Lipoprotein glomerulopathy is characterized by nephritic syndrome glomerular protein thrombi and lipid abnormalities, particularly with an elevated level of plasma apoprotein E (apoE).There are no efficiency way to treat lipoprotein glomerulopathy. We firstly successfully treat 2 patients by protein A immunoadsorption with remarkable decreased urine protein and reduction of lipoprotein thrombi on repeated renal biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. A new diagnosis of lipoprotein glomerulopathy proved by histology and serology
2. Age 15~60 years, sex free

Exclusion Criteria:

1. Serum creatinine > 500 umol/l
2. Severe viral infection(HBV, HCV, CMV) within 3 months of first randomization or known HIV infection
3. Congenital or acquired immunodeficiency
4. Patients with severe infection or central nervous system symptoms
5. Immediately life-threatening organ manifestations (e.g. lung haemorrhage or massive gastro-intestinal bleeding, heart failure due to pericarditis or myocarditis, liver dysfunction measured on at least 2 separate occasion)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2000-01; Primary Completion 2002-03 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of immunoadsorption in the treatment of lipoprotein glomerulopathy. | 3 months

SECONDARY OUTCOMES:
To assess the safety of immunoadsorption in the treatment of lipoprotein glomerulopathy. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-hong Liu, M.D., Principal Investigator — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China